CLINICAL TRIAL: NCT00655278
Title: Phase II Efficacy and Safety of Taro Pharmaceuticals' Pro-Drug T2000 (1,3-dimethoxymethyl-5,5-diphenyl-barbituric Acid) in Patients With Essential Tremor: An Open-Label Dose Continuation Study
Brief Title: T2000 in Essential Tremor - Open Label Continuation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2000-0639
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-11

CONDITIONS: Essential Tremor
Keywords: Movement Disorder
MeSH Terms: conditions — Essential Tremor; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): T2000 at 600-1000 mg daily
  Interventions: Drug: T2000

INTERVENTIONS:
Drug: T2000 — T2000 at previous most effective, well-tolerated dose (600-1000mg daily)

SUMMARY:
This study will evaluate the safety and efficacy of T2000 when used to treat patients with moderate to severe essential tremor over an 18 month period.

DETAILED DESCRIPTION:
Essential tremor (ET) is a common form of involuntary shaking not related to Parkinson's disease. The medications that are currently used to treat ET work in a small proportion of patients and provide only partial improvement in symptoms. Use of these current medications is also limited by side-effects in many patients.

T2000 is a medication currently under development for the treatment of essential tremor. Although T2000 is a new medication, it belongs to a class of medications that has been used for many years for the treatment of a variety of medical conditions. In previous studies, T2000 appeared to be effective in controlling symptoms of ET and some patients with severe ET had major improvements in tremor. In some patients T2000 was well tolerated for periods up to 5 months and the minimal side-effects seen were those that would be expected for medications in this class.

The current study will evaluate the safety and efficacy of T2000 in patients with moderate to severe essential tremor. Patients will receive doses of T2000 beginning at 600 mg a day, followed by 800 mg a day and up to 1000 mg a day. The total duration of treatment will be 18 months. Patient's tremor and neurological examination will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Patients will be enrolled following completion of a dose escalation trial (such as T2000-0533)

* Confirmed essential tremor by NIH criteria
* Significant functional activity limitation due to ET
* Patients who have failed, are inadequately treated or cannot tolerate alternative treatments for ET as well as treatment naïve patients who have considered but declined alternative treatment

Exclusion Criteria:

* Patients adequately controlled without side effects on a current ET treatment
* Pregnant patients or patients who may become pregnant during the study
* Patients with other medical conditions that may cause tremor, such as Parkinson's disease or active hyperthyroidism
* Patients taking medications that might produce tremor or interfere with the evaluation of tremor such as CNS-stimulants or beta-blockers
* Patients who must take medications that alter liver metabolism as well as patients with liver disease or coagulation disorders
* Patients with seizure disorders
* Patients with a history of allergy or hypersensitivity reaction to barbiturates or other related medications, such as phenobarbital or phenytoin
* Patient with significant general medical or clinical laboratory abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-08; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Effect of treatment on tremor will be measured by a tremor scale as well as by assessment of functional activity with specific tasks. | Up to 18 months

SECONDARY OUTCOMES:
Safety parameters including neurological examination, blood tests and EKG will be monitored throughout the treatment period and during withdrawal of the medication. | Up to 18 months

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Investigator Site, London, Ontario
  - Investigator Site, Ottawa, Ontario
  - Investigator Site, Toronto, Ontario

REFERENCES:
- [Background] Melmed C, Moros D, Rutman H. Treatment of essential tremor with the barbiturate T2000 (1,3-dimethoxymethyl-5,5-diphenyl-barbituric acid). Mov Disord. 2007 Apr 15;22(5):723-7. doi: 10.1002/mds.21321. PMID 17265458